CLINICAL TRIAL: NCT02399228
Title: An Open-Label, Proof of Concept, Efficacy, Safety and Tolerability Trial of a Botanical Drug Containing East Indian Sandalwood Oil (EISO) for the Prevention and Treatment of Oral Mucositis Induced by Radiation Therapy
Brief Title: A Trial of a Botanical Drug Containing East Indian Sandalwood Oil (EISO) for the Treatment of Oral Mucositis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santalis Pharmaceuticals, Inc. (Industry)
Collaborators: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SAN005-01
Record Dates: First submitted 2015-03-17; First posted 2015-03-26 (Estimated); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Oral Mucositis
Keywords: radiation therapy; chemotherapy; head and neck cancer
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 0.25% EISO Mouth Rinse (Experimental): A mouth rinse containing 0.25% East Indian sandalwood oil (EISO), a candidate botanical drug substance. The rinse will be used three times a day for up to ten weeks. The material will not be ingested but used to "swish, gargle and spit".
  Interventions: Drug: 0.25% EISO mouth rinse

INTERVENTIONS:
Drug: 0.25% EISO mouth rinse — A mouth rinse to be used three times a day during the course of radiation and/or chemotherapy to prevent or minimize oral mucositis
  Other Names: East Indian sandalwood oil, Albuterpenoids

SUMMARY:
The initial proposed clinical study will be conducted in adult head and neck cancer subjects. This will be an open-labeled, proof of concept trial to evaluate the efficacy, safety and tolerability of EISO in a form of oral rinse as adjunctive therapy to standard of care. Santalis believes that the proposed study is a prudent and appropriate approach to investigate the potential of their product to prevent or improve oral mucositis symptoms commonly seen in subjects undergoing radiotherapy with or without chemotherapy.

DETAILED DESCRIPTION:
The objectives of this proof of concept trial are: to evaluate the efficacy, safety and tolerability of SAN005 when administered to adults for the prevention and treatment of radiation induced oral mucositis.

Subjects will be instructed on the administration of study medication thrice daily till oral mucositis resolves. Subjects will return to the clinic once a week while receiving radiation and then once every two weeks once their radiation has been completed and then until their mucositis has resolved for the Final Study Visit.

Preliminary Efficacy Evaluation will be the severity of pain rated by the Numeric Pain Rating Scale (NRPS) and mucositis grade by Radiation Therapy Oncology Group (RTOG) criteria at Visit 7 (Day 36). Additional secondary efficacy evaluations will include the severity of pain rated by the NRPS and mucositis grade by RTOG criteria at each study visit, frequency of the percutaneous endoscopic gastrostomy (PEG) tube for feeding during the duration of treatment and weight loss from baseline through Visit 5 and 7. The time of mucositis onset and duration will also be used in assessing efficacy. Additional secondary and exploratory endpoints will be outlined in the statistical analysis plan. The overall efficacy is determined by comparing the data to historical controls. Safety will be assessed by evaluating adverse events (AEs) with respect to severity, duration, and relationship to study drug. In addition, tolerability evaluations will be performed at each study visit.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with head and neck cancer involving the oropharynx or oral cavity, who are expected to undergo high dose radiation therapy (i.e., ≥ 60 Gy) that typically results in oral mucositis, with or without concurrent chemotherapy or biologic targeted therapy.
2. At least 18 years of age
3. Estimated survival of at least 6 months.
4. No prior radiation therapy to the head and neck area, and no chemotherapy within the last year except for induction chemotherapy delivered (or to be delivered) prior to the current course of radiation therapy
5. Female subjects of child-bearing potential must agree to use an adequate form of contraceptive (e.g., hormonal, barrier method or abstinence) prior to study entry and for the duration of the trial.
6. Are willing to refrain from using other treatments for oral mucositis until they consult with the study investigator(s).
7. Are able to give written informed consent in a manner approved by the Institutional Review Board and comply with the requirements of the study.

Exclusion Criteria:

1. Have preexisting mucositis from other causes.
2. Are immunosuppressed or in chronic use of immunosuppressive drugs.
3. Have a known sensitivity to any of the constituents of the test product including sensitivities to sandalwood oil, fragrances or any member of the Compositae family of vascular plants (e.g., sunflowers, daisies, dahlias, etc.).
4. Eastern Cooperative Oncology Group (ECOG) performance status > 3
5. Unwilling or unable to follow the protocol requirements.
6. Have any condition that in the opinion of the investigator would confound the efficacy, safety and tolerability assessments, such as oral thrush.
7. Have participated in any clinical trial in the previous 30 days.
8. Are pregnant, breastfeeding, or unwilling to practice an acceptable form of birth control during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-10-04 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Castella, PhD, Study Director — Santalis Pharmaceuticals
Locations (1):
- UTHSCSA Cancer Therapy and Research Center (CTRC), San Antonio, Texas, United States

REFERENCES:
- [Background] Rosenthal DI, Trotti A. Strategies for managing radiation-induced mucositis in head and neck cancer. Semin Radiat Oncol. 2009 Jan;19(1):29-34. doi: 10.1016/j.semradonc.2008.09.006. PMID 19028343
- [Background] Singh CU NJ, inventors. : Derivatives of sandalwood oil and santalols for treating cold sores and herpes. . US patent application publication US2008/0058413 A1. 06 2008

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.25% EISO Mouth Rinse
Started | 13
Completed | 7
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | 0.25% EISO Mouth Rinse
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 3
Age, Continuous [Mean (Full Range); unit: years] | 55.4 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Patients Achieving Less Than or Equal to "2" RTOG Score At Visit 9
Description: The Radiation Therapy Oncology Group (RTOG) is the measure of anatomical changes associated with oral mucositis. Patients scores will be compared to historical data of patient progression.
  RTOG Scoring Criteria- Grade 0(none)- No change over baseline Grade 1(mild)- Irritation, may experience slight pain, not requiring analgesic Grade 2(moderate)- Patchy mucositis that may produce inflammatory serosanguinitis discharge; may experience moderate pain requiring analgesia Grade 3(severe) -Confluent, fibrinous mucositis, may include severe pain requiring narcotic Grade 4(life-threatening)-Ulceration, hemorrhage, or necrosis
Time Frame: Up to ten (10) weeks
Population: Not all subjects analyzed at visit 9 completed the trial. Therefore, the number of completed subjects (7) is less than the number of subjects analyzed for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% EISO Mouth Rinse
Number analyzed (Participants) | 7
Participants | 7

2. Secondary Outcome: Subject Self Reporting Burning or Irritation
Description: Calculated by the number and percentage of subjects self reporting irritation of grade 1 (mild) or higher.
Time Frame: Up to ten (10) weeks
Population: All subjects who reported tolerability at any point during the study were analyzed
Measure: Count of Participants; unit: Participants
Arm/Group | 0.25% EISO Mouth Rinse
Number analyzed (Participants) | 13
Participants
  None | 4
  Mild | 4
  Moderate | 3
  Severe | 2

3. Secondary Outcome: NRPS (Numerical Rating Pain Scale)
Description: Severity of pain in the oral cavity/oropharynx was measured using the numerical rating pain scale (NRPS) at each study visit. The NRPS is an 11-point scale from 0-10:
  0 = No pain 10 = The most intense pain imaginable.
Time Frame: Up to ten (10) weeks
Population: ITT (Intention-to-treat)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 0.25% EISO Mouth Rinse
Number analyzed (Participants) | 13
score on a scale | 3.875 (2.75)

4. Other Pre Specified Outcome: Safety Will be Assessed Based on the Frequency and Severity of Adverse Events.
Description: Adverse Events (AEs) will be assessed in accordance the Common Terminology Criteria for Adverse Events (CTCAE). The number of patients experiencing adverse events possibly, or probably related to the study product will be reported.
  Possibly related: A clinical event, including laboratory test abnormality (if applicable), with a reasonable time sequence to administration of the drug, but which could also be explained by concurrent disease or other drugs or chemicals.
  Probably related: A clinical event, including laboratory test abnormality (if applicable), with a reasonable time sequence to administration of the drug, unlikely to be attributed to concurrent disease or other drugs or chemicals, and which follows a clinically reasonable response on withdrawal.
Time Frame: [ Time Frame: Up to ten (10) weeks ]
Population: Only 4 patients reported adverse events possibly or probably related to the study product.
Measure: Number; unit: participants
Arm/Group | 0.25% EISO Mouth Rinse
Number analyzed (Participants) | 13
participants
  Nausea (Mild) | 2
  Vomiting (Mild) | 2

ADVERSE EVENTS:
Time Frame: Over the course of the treatment (up to 10 weeks), which was while the patients were undergoing radiotherapy and chemo.
Description: Adverse events were solicited from subjects through clinic visits and captured on daily diaries
Arm/Group | 0.25% EISO Mouth Rinse
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.25% EISO Mouth Rinse (N=13)
Nausea (Gastrointestinal disorders) | 6 (6)
Vomiting Grade 1 (Gastrointestinal disorders) | 3 (3)
Dysgeusia (General disorders) | 6 (6)
Dry Mouth (General disorders) | 5 (5)
Fatigue (General disorders) | 5 (5)
Dermatitis Radiation (Skin and subcutaneous tissue disorders) | 4 (4)
Weight Loss (General disorders) | 4 (4)
Dysphagia (General disorders) | 3 (3)
Insomnia (General disorders) | 3 (3)
Mucositis (Skin and subcutaneous tissue disorders) | 3 (3)
Anemia (Metabolism and nutrition disorders) | 2 (2)
Cough (General disorders) | 2 (2)
Creatinine Increased (Renal and urinary disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Ear Pain (Ear and labyrinth disorders) | 2 (2)
Hypoalbuminemia (General disorders) | 2 (2)
Hypocalcemia (Renal and urinary disorders) | 2 (2)
Hypomagnesemia (General disorders) | 2 (2)
Hyponatremia (General disorders) | 2 (2)
Lymphocyte count decreased (Immune system disorders) | 2 (2)
Mucosal Infection (Immune system disorders) | 2 (2)
Oral Pain (General disorders) | 2 (2)
Sore Throat (General disorders) | 2 (2)
White Blood Cell Decreased (Immune system disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Constipation (General disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Epistaxis (General disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Hypokalemia (General disorders) | 1 (1)
Memory Impairment (Psychiatric disorders) | 1 (1)
Neutrophil Count Decreased (Immune system disorders) | 1 (1)
Otitis Externa (Eye disorders) | 1 (1)
Otitis Media (Eye disorders) | 1 (1)
Platelet Count Decreased (Immune system disorders) | 1 (1)
Tumor Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-01-27): https://cdn.clinicaltrials.gov/large-docs/28/NCT02399228/Prot_SAP_000.pdf
  • Informed Consent Form (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/28/NCT02399228/ICF_001.pdf